CLINICAL TRIAL: NCT00369564
Title: Glutamic Acid to Decrease Vincristine Toxicity in Children With Cancer
Brief Title: Glutamic Acid in Reducing Nerve Damage Caused by Vincristine in Young Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SCUSF 0402; SCUSF 0402 (Other: SunCoast CCOP Research Base); ACCL 0731 (Other: Children's Oncology Group); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2018-09

CONDITIONS: Kidney Cancer; Leukemia; Lymphoma; Neurotoxicity; Peripheral Neuropathy; Sarcoma
Keywords: neurotoxicity; peripheral neuropathy; stage I Wilms tumor; stage II Wilms tumor; stage III Wilms tumor; stage IV Wilms tumor; stage V Wilms tumor; previously untreated childhood rhabdomyosarcoma; childhood grade III lymphomatoid granulomatosis; childhood diffuse large cell lymphoma; childhood immunoblastic large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; childhood Burkitt lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma; untreated childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Kidney Neoplasms; Leukemia; Lymphoma; Neurotoxicity Syndromes; Peripheral Nervous System Diseases; Sarcoma; Wilms Tumor; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma | interventions — Glutamic Acid; glutamic acid diethyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I Glutamic Acid (Experimental): Patients receive oral glutamic acid 3 times daily beginning prior to the first dose of vincristine and continuing through week 5 (stratum 2) or week 10 (stratum 1).
  Interventions: Drug: glutamic acid
- Arm II Placebo (Placebo Comparator): Patients receive oral placebo 3 times daily beginning prior to the first dose of vincristine and continuing through week 5 (stratum 2) or week 10 (stratum 1).
  Interventions: Other: placebo

INTERVENTIONS:
Drug: glutamic acid — Given orally 3 times daily
  Other Names: l-glutamic acid hydrochloride
  Arms: Arm I Glutamic Acid
Other: placebo — Given orally 3 times daily
  Arms: Arm II Placebo

SUMMARY:
RATIONALE: Glutamic acid may help lessen or prevent nerve damage caused by vincristine. It is not yet known whether glutamic acid is more effective than a placebo in preventing nerve damage in patients receiving vincristine for Wilms' tumor, rhabdomyosarcoma, acute lymphoblastic leukemia, or non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying glutamic acid to see how well it works compared to a placebo in reducing nerve damage caused by vincristine in young patients receiving vincristine for Wilms' tumor, rhabdomyosarcoma, acute lymphoblastic leukemia, or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of glutamic acid vs placebo, in terms of decreasing neurotoxicity as measured by a scored neurologic examination, in young patients undergoing vincristine-containing treatment for Wilms' tumor, rhabdomyosarcoma, acute lymphoblastic leukemia, or non-Hodgkin's lymphoma.

Secondary

* Compare the frequency and types of neurotoxicity observed in patients treated with glutamic acid versus placebo.
* Determine if a greater proportion of patients receiving glutamic acid are able to receive 100% of their scheduled doses of vincristine versus those not treated with glutamic acid.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease and duration of planned vincristine-containing treatment (Wilms' tumor or rhabdomyosarcoma with treatment planned for ≥ 9 consecutive weeks [stratum 1] vs acute lymphoblastic leukemia or non-Hodgkin's lymphoma with treatment planned for ≥ 4 consecutive weeks [stratum 2]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral glutamic acid 3 times daily beginning prior to the first dose of vincristine and continuing through week 5 (stratum 2) for a total of 4 doses of vincristine or week 10 (stratum 1) for a total of 9 doses of vincristine.
* Arm II: Patients receive oral placebo 3 times daily beginning prior to the first dose of vincristine and continuing through week 5 (stratum 2) for a total of 4 doses of vincristine or week 10 (stratum 1) for a total of 9 doses of vincristine.

All patients undergo neurologic examination at baseline and at 5 weeks. Patients in stratum 1 also undergo additional neurologic examination at week 10.

PROJECTED ACCRUAL: A total of 250 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients ≥ 3 and < 21 years of age at the time of study registration.
* Patients newly diagnosed with Wilm's tumor and scheduled to receive at least 9 consecutive weeks of chemotherapy with a vincristine-containing regimen.
* Patients newly diagnosed with rhabdomyosarcoma and scheduled to receive at least 9 consecutive weeks of chemotherapy with a vincristine-containing regimen.
* Patients newly diagnosed with ALL and scheduled to receive 4 consecutive weeks of chemotherapy with a vincristine-containing regimen with accompanying steroid therapy.
* Patients newly diagnosed with Non- Hodgkins Lymphoma (NHL) and scheduled to receive 4 consecutive weeks of chemotherapy with a vincristine-containing regimen with accompanying steroid therapy.
* Patients with no underlying neuromuscular disease or peripheral neuropathy

EXCLUSION CRITERIA:

* Abnormal baseline peripheral neurologic exam (i.e. or peripheral neuropathy)
* Patients with:
* seizure disorders
* primary intracranial malignancy
* family history of Charcot Marie Tooth Disease
* a recent history of GuillianBarré26
* Patients receiving concomitant itraconazole are at risk for increased vincristine toxicity and therefore are ineligible.
* Patients who are regularly using laxatives or stool softeners for constipation at the time of enrollment are not eligible to participate in the study. Likewise, since prevention of neuro-constipation will be evaluated, patients with an ongoing history of constipation that has required frequent use of laxatives or stool softeners should not be enrolled.
* Patients should not be scheduled to receive laxatives or stool softeners prophylactically to prevent constipation, as the prevention of neuro-constipation will be evaluated in this study; however, when patients show signs of developing constipation while on chemotherapy, as determined by the treating physician, they may be treated with laxatives or stool softeners at the clinician's discretion. Use of laxatives or stool softeners will be documented on the concomitant medication log.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2007-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Bradfield, MD, Study Chair — Nemours Children's Clinic; Eric Sandler, MD, Study Chair — Nemours Children's Clinic; David R. Freyer, DO, MS, Study Chair — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I Glutamic Acid: Patients receive oral l-glutamic acid hydrocloride 3 times daily beginning prior to the first dose of vincristine and continuing through week 5 (stratum 2) or week 10 (stratum 1). Patients with a body surface area (BSA) less than 1.0 m^2 will receive a total of 750 mg/day of oral glutamic acid . Patients with a body surface area (BSA) greater or equal to1.0 m^2 will receive a total of 1500 mg/day of oral glutamic acid .
- Arm II Placebo: Patients receive oral placebo 3 times daily beginning prior to the first dose of vincristine and continuing through week 5 (stratum 2) or week 10 (stratum 1). Placebo capsules are identical in appearance to the active oral glutamic acid capsules but instead each capsule contains 324 mg of microcrystalline cellulose as a filler, 3 mg of magnesium stearate as a lubricant and 3 mg silicone dioxide as a drying agent for a total fill weight of 330 mg. The manufacturer has certified that the placebo contains no active agent.
  Patients with a body surface area (BSA) less than 1.0 m^2 will receive a 1 capsule of placebo 3 times daily (total 3 capsules daily). Patients with a body surface area (BSA) greater or equal to1.0 m^2 will receive a 2 placebo capsules 3 times daily (total 6 capsules daily). .
Period: Overall Study
Arm/Group | Arm I Glutamic Acid | Arm II Placebo
Started | 127 | 123
Completed | 84 | 100
Not Completed | 43 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Glutamic Acid | Arm II Placebo | Total
Number analyzed (Participants) | 127 | 123 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 123 | 117 | 240
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (4.8) | 8.6 (4.9) | 8.6 (4.9)
Sex/Gender, Customized [Number; unit: participants] — One subject did not report gender information.
  participants
    Gender- Female | 46 | 53 | 99
    Gender- Male | 81 | 69 | 150
    Gender Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 127 | 123 | 250

OUTCOME MEASURES:

1. Primary Outcome: Neurotoxicity as Measured by a Scored Neurologic Examination at Baseline, 5 Weeks, and 10 Weeks (if Applicable)
Description: A neurological exam will be completed at baseline and at study week 5 for both strata. An additional exam at week 10 will be done for patients in Stratum 1. Additional exams will be done at any time if the treating oncologist deems it clinically necessary . Neurotoxicity will be scored using a standardized neurological exam form developed for the study that is based on the Modified "Balis" Pediatric Scale of Peripheral Neuropathies. Treatment groups will be compared with respect to the proportion experiencing a grade 2 or higher toxicity from the following list of neurologic toxicities captured on the Neurologic Exam Form including sensory neuropathy, motor neuropathy, laryngeal nerve, constipation/neuro-constipation, jaw pain, or other specified abnormalities noted by the attending physician. Percentage of patients with one or more Grade 2 or higher noted neurotoxicity symptoms on any item in the Balis scale will compared between arms.
Time Frame: 10 weeks
Population: Patients reporting baseline and post-baseline observation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I Glutamic Acid | Arm II Placebo
Number analyzed (Participants) | 97 | 107
percentage of participants | 26 (4.4) [18 to 37] | 34 (4.5) [23 to 41]

2. Secondary Outcome: Number of Participants With Neurotoxicity Observed
Description: Number of participants with neurotoxicity observed treated with l-glutamic acid hydrochloride as compared to the number of participants with neurotoxicity observed in the placebo control group
Time Frame: 10 weeks
Population: Stratum 2 with a >= grade 2 neurotoxicity
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Glutamic Acid | Arm II Placebo
Number analyzed (Participants) | 79 | 88
Participants | 21 | 25

3. Secondary Outcome: Ability to Receive All Scheduled Doses of Vincristine
Description: We will determine if a greater proportion of patients receiving l-glutamic acid hydrochloride are able to receive 100% of their scheduled doses of vincristine as compared to those in the placebo control group
Time Frame: 10 weeks
Population: Number in stratum 1 and stratum 2 that completed
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Glutamic Acid | Arm II Placebo
Number analyzed (Participants) | 127 | 123
Participants | 84 | 100

4. Secondary Outcome: Types of Neurotoxicities
Description: Types of neurotoxicities reported. Each patient was only counted once for each type of neurotoxicity, but a patient could be counted in more than 1 type of neurotoxicity. For example, if a patient experienced constipation 3 times, they are included once for constipation. If a patient experienced sensory changes and motor changes, they are included once for sensory changes and once for motor changes.
Time Frame: 10 Weeks
Population: Participants who returned a post baseline Neurotox Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I Glutamic Acid | Arm II Placebo
Number analyzed (Participants) | 127 | 123
Participants
  Constipation: number analyzed (Participants) | 97 | 107
  Constipation | 11 | 14
  Sensory Changes: number analyzed (Participants) | 97 | 107
  Sensory Changes | 11 | 13
  Motor Changes: number analyzed (Participants) | 97 | 107
  Motor Changes | 10 | 13
  Jaw Pain: number analyzed (Participants) | 97 | 107
  Jaw Pain | 4 | 2
  Laryngeal Nerve Dysfunction: number analyzed (Participants) | 97 | 107
  Laryngeal Nerve Dysfunction | 2 | 1

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: Subjects and parents completed daily study medication logs and noted any adverse events or symptoms. Site personnel reviewed study medication logs with subjects to assess for adverse events and completed an in-person neurological exam and chemistry profile at weeks 5 and 10 to assess for adverse events. Adverse events reviewed by independent DSMB.
Arm/Group | Arm I Glutamic Acid | Arm II Placebo
Serious Adverse Events (participants affected / at risk) | 9/127 | 6/123
Other Adverse Events (participants affected / at risk) | 16/127 | 5/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Glutamic Acid (N=127) | Arm II Placebo (N=123)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (General disorders) | 1 (1) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0)
Febrile neutropenia (Infections and infestations) | 1 (1) | 1 (2)
Infection-Other (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC (Infections and infestations) | 1 (2) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Leukoencephalopathy (radiographic findings) (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vascular - Other (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I Glutamic Acid (N=127) | Arm II Placebo (N=123)
Vomiting (Gastrointestinal disorders) | 9 (10) | 3 (3)
Pain (General disorders) | 7 (7) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No